CLINICAL TRIAL: NCT01188278
Title: Treatment With Second Generation TYROSINE KINASE INHIBITORS (2G TKI) Post Imatinib Failure: Factors Predicting Response and Predictive Value of Response
Brief Title: Treatment With Second Generation Tyrosine Kinase Inhibitors (2G TKI) Post Imatinib Failure Survey
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-291
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2013-10

CONDITIONS: Leukemia, Myeloid, Chronic-Phase (CML-CP)
MeSH Terms: conditions — Leukemia | interventions — Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in CP-CML treated with 2G TKI: Patients in CP-CML treated with 2G TKI (nilotinib or dasatinib) post imatinib failure
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Drug being observed but not provided
  Other Names: Dasatinib; Nilotinob

SUMMARY:
The purpose of this study is to determine predictive value of Hammersmith score on Complete Cytogenetic Response (CCyR).

DETAILED DESCRIPTION:
Historic cohort prolonged by a 12-month follow-up period.

Prospective: look forward using periodic observations collected predominantly following subject enrollment: one year of follow up of patients with CP-CML alive at the time of the study.

Retrospective: look back using observations collected predominantly prior to subject selection and enrollment : historical data of patients with CP-CML initiated with a 2G TKIs post-imatinib failure (resistance or intolerance) between 1-Jan-2005 and 30-June-2009.

The inclusion of a historical cohort will allow a rapid enrollment of a large number of patients of this rare pathology, while the prospective follow up of this cohort would allow long term data to be obtained, including the assessment of the impact on survival and appreciate the patient's quality of life (QoL), compliance and satisfaction.

ELIGIBILITY:
Patients with Additional Chromosomal Anomalies (ACA) are accepted to be in CP. Patients enrolled in open-label clinical trials or other observational trials are also allowed (unless explicitly prohibited by the trial).

This trial does not prohibit participation in other observational trials.

Inclusion Criteria:

* Patients diagnosed with CP-CML. (ACA) are allowed
* Age >18 years old
* Prior treatment with imatinib monotherapy as first line treatment, to which the patient is deemed resistant or intolerant.Patients treated by INF and/or AraC prior (but not concomitant) to imatinib are eligible.
* Initiated with a 2G TKIs post-imatinib failure (resistance or intolerance) between 1-Jan-2005 and 30-Jun-2009.

Exclusion Criteria:

* Patients in (or with history of) accelerated or blastic phase CML
* Patients treated by allogeneic stem cell transplantation.
* Any other CML treatment except for INF and/or AraC,and a short period of Hydroxyurea or Anagrelide prior to imatinib.
* Patients treated with 2G TKI for reasons other than imatinib failure.
* Patients with no historical data (e.g. possibility of Sokal Score calculation) available.
* Patients participating in clinical or observational trials which explicitly prohibit enrollment in non interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematology centers (hospitals) which have necessary historical data available
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Predictive value of Hammersmith score on Complete Cytogenetic Response (CCyR) | CCyR at 6 month of 2GTKI treatment
  The purpose of this study is to determine predictive value of Hammersmith score on Complete Cytogenetic Response (CCyR), as assessed by the following:
  * Distribution of patients according to Hammersmith score levels
  * Characterization of association between Hammersmith score and occurrence of CCyR
  * Assessment of capacity of Hammersmith score to predict CCyR, using diagnostic test assessment methods.
  This score is measured at the time of imatinib failure.

SECONDARY OUTCOMES:
Predictive value of Hammersmith score on Major Molecular Response (MMR) | MMR at 3 month of 2GTKI treatment
  The purpose of this study is to determine predictive value of Hammersmith score on Major Molecular Response(MMR), as assessed by the following:
  * Distribution of patients according to Hammersmith score levels
  * Characterization of association between Hammersmith score and occurrence of MMR
  * Assessment of capacity of Hammersmith score to predict MMR, using diagnostic test assessment methods.
  This score is measured at the time of imatinib failure.
Predictive factors of Overall survival (including Hammersmith score, MMR at 3 months and CCyR at 6 months of 2G TKI treatment together with patients, disease and treatment characteristics) | From switch to 2G TKI between 01Jan2005 and 30Jun2009 to 31Oct2011 if alive or to the death
Predictive value of Hammersmith score compared to other factors | From switch to 2G TKI between 01Jan2005 and 30Jun2009 to 31Oct2011 if alive or to the death
  imatinib treatment duration, mutations at time of failure, best response to imatinib, time between imatinib failure & initiation of 2G TKI on the response to 2G TKI & on the survival end points (Overall Survival (OS)& Progression Free Survival (PFS)).
Patients populations (socio-demographic data, medical history, disease history, co morbidities treated with 2G TKI | When occurs the switch from Imatinib to 2G TKI between 01Jan2005 and 30Jun2009
Patients' satisfaction, Quality of life & compliance to treatment in patients treated with 2G TKIs | For all alive patients treated with 2G TKI during the enrolment period (Jun2010 to Oct2010)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm